CLINICAL TRIAL: NCT04059016
Title: NIDA CTN Protocol 0090 Innovatively Increasing PCP Prescribing of Buprenorphine: Measurement Based Care and Integrated Electronic Solution (MBC4OUD)
Brief Title: Innovatively Increasing PCP Prescribing of Buprenorphine: Measurement Based Care and Integrated Electronic Solution
Acronym: MBC4OUD
Status: Completed | Type: Observational
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Madhukar H. Trivedi, MD, Professor, University of Texas Southwestern Medical Center
Other Study IDs: STU-2019-0743; UG1DA020024 (NIH)
Record Dates: First submitted 2019-07-16; First posted 2019-08-16 (Actual); Last update posted 2024-06-18 (Actual); Status verified 2024-06

CONDITIONS: Opioid Abuse and Addiction
Keywords: opioid use disorder; buprenorphine waiver training; VitalSign6; measurement based care; primary care
MeSH Terms: conditions — Opioid-Related Disorders; Behavior, Addictive

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: MBC4OUD — This computer software program consists of patient-completed self reports for screening and diagnosis of opioid use disorder among primary care patients and provides web-based clinical decision support to primary care providers for provision of pharmacotherapy for opioid use disorder.

SUMMARY:
The objective of this observational feasibility project is to assess the feasibility and acceptability of universal screening and measurement based care for opioid use disorder (OUD) utilizing a computer software program in a network of primary care clinics currently utilizing this software for screening and measurement based care (MBC) for the treatment of depression. The primary objective of this project is to evaluate the feasibility of screening and MBC for OUD in our partner primary care clinics. The secondary objective of this project is to evaluate the acceptability of universal screening and measurement based care of OUD, including the barriers and facilitators of screening for OUD and providing buprenorphine treatment in primary care, changes in provider knowledge and beliefs regarding diagnosis and treatment of OUD, and treatment program outcomes.

DETAILED DESCRIPTION:
This is an observational feasibility project evaluating the impact of universal screening and enhanced access to care for patients with opioid use disorder via development and implementation of web-based software program that provides clinical decision support to primary care providers for the diagnosis and treatment of opioid use disorder (OUD) with buprenorphine. The key facets of measurement based care (MBC) for OUD will be supported by the software: (1) screening instrument used for all patients, (2) diagnostic instrument for patients who screen positive, and (3) buprenorphine treatment algorithm for those with diagnosed OUD. The MBC for OUD software will be offered to clinics in the University of Texas Southwestern Medical Center (UTSW) North Texas Community Based Primary Care Network. Clinics in the Network currently utilize VitalSign6, a software program that implements universal screening for depressive symptoms and provides electronic clinical decision support for measurement based care (MBC) for major depression. The VitalSign6 team provides training on how to clinically diagnose and manage major depression, training on the software, and expert clinical support during implementation.

Clinics in the Network will be offered the opportunity to utilize the newly developed VS6 OUD diagnosis and treatment module. Network clinics that take part in this project will be provided training in the diagnosis and management of OUD and federally-mandated training in the use of buprenorphine for OUD. The primary outcome will be the number of primary care providers trained to prescribe buprenorphine for OUD (i.e., complete waiver training). The providers and staff at clinics who choose to utilize the newly developed VS6 OUD module (i.e., MBC4OUD) will be invited to participate in a research project assessing acceptability of the diagnosis and treatment of OUD in primary care.. Focus groups will be utilized to assess stakeholder barriers to implementation of buprenorphine treatment for OUD and strategies for overcoming these barriers. Providers at clinics taking part in the project will be surveyed regarding their beliefs and comfort level with OUD diagnosis and treatment at 3 time-points: pre-training, post-training (i.e., prior to software dissemination to the clinic when the observation period begins), and at the end of the observation period. All data from providers will be collected anonymously. De-identified patient level data will be analyzed for the purpose of program evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Providers and clinical staff from UTSW clinics currently utilizing the VitalSign6 software program

Exclusion Criteria:

-

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Providers and clinical staff from clinics in the University of Texas Southwestern Medical Center (UTSW) North Texas Community Based Primary Care Network that currently utilize VitalSign6, a software program that implements universal screening for depressive symptoms and provides electronic clinical decision support for measurement based care (MBC) for major depression.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2024-05-02 (Actual); Study Completion 2024-05-02 (Actual)

PRIMARY OUTCOMES:
% of primary care providers completing buprenorphine waiver training | 3 months
  The number of primary care providers who complete buprenorphine waiver training divided by the divided by the number of providers who indicate a desire/willingness to be trained will be computed.

SECONDARY OUTCOMES:
Clinic Interest Rate | 3 months
  The number of Network clinics who accept the OUD module divided by the number of clinics that were approached.
Provider Buprenorphine Waiver Training Completion Rate | 3 months
  The number of providers in Network clinics who complete buprenorphine waiver training divided by the number of providers who indicated desire/willingness to complete the buprenorphine waiver training.
OUD Module Training Completion Rate | 3 months
  The number of providers who complete the VS6 OUD module training divided by the number of providers who indicated desire/willingness to complete the VS6 OUD module training.
Buprenorphine Treatment Acceptability Scale | 3 months
  The Buprenorphine Treatment Acceptability Scale has been created by the investigators for this study. It is a 29-item self report measure. Items 1-27 are assessed on 1-5 Likert scale, with 1=strongly disagree and 5=strongly agree. Items 28 and 29 are scored on a scale of 0-100, with higher scores indicating greater confidence. Items on the scale assess provider motivation for providing treatment for opioid use disorder, provider self-efficacy for the treatment of opioid use disorder, and challenges faced by providers in treating opioid use disorder.

CONTACTS AND LOCATIONS:
Overall Officials: Madhukar H Trivedi, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- University of Texas Southwestern Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be transmitted to the NIDA central data repository as requested by NIDA. The data management team will conduct final data quality assurance checks and "lock" the database from further modification. The final analysis dataset will be returned to NIDA, as requested, for storage and archive.
Supporting Information: Study Protocol

REFERENCES:
- [Derived] Dela Cruz AM, Karns-Wright T, Kahalnik F, Walker R, Lanham HJ, Potter JS, Trivedi MH. Stigma towards opioid use disorder in primary care remain a barrier to integrating software-based measurement based care. BMC Psychiatry. 2023 Oct 24;23(1):776. doi: 10.1186/s12888-023-05267-w. PMID 37875835
- [Derived] Dela Cruz AM, Walker R, Pipes R, Wakhlu S, Trivedi MH. Creation of an algorithm for clinical decision support for treatment of opioid use disorder with buprenorphine in primary care. Addict Sci Clin Pract. 2021 Feb 19;16(1):12. doi: 10.1186/s13722-021-00222-0. PMID 33608060